CLINICAL TRIAL: NCT06866327
Title: Feasibility and Acceptability of Music Training Programs Among Older Adults Living with Mild Cognitive Impairment: a Pilot Randomized Controlled Trial
Brief Title: Music for the Mind Study
Acronym: M4M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Eastman Performing Arts Medicine Center (Unknown); University of Rochester Aging Institute (Unknown); University of Rochester School of Nursing (Unknown)
Responsible Party: Principal Investigator, Kathi Heffner, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00010048
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment (MCI); Memory Disorders, Age Related; Memory Decline
Keywords: music; memory; mood; emotion; well-being
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Piano lessons (Experimental): Introduction to piano playing, including instruction and practice in note reading, finger positions, and song playing.
  Interventions: Behavioral: Piano lessons
- Music lessons (Active Comparator): Introduction to varied instrument playing, music singing, and music appreciation.
  Interventions: Behavioral: Music Lessons

INTERVENTIONS:
Behavioral: Piano lessons — The program consists of 12-weekly piano lessons, alternating small group lessons and individual lessons each week. Individual lessons reinforce and help personalize what is instructed during group lessons. Lessons are tailored to help older adults with memory challenges learn note reading, finger positioning, and song playing. Participants are asked to practice at home in between lessons for 10 minutes per day, 5 times per week, with a keyboard and bench provided.
  Arms: Piano lessons
Behavioral: Music Lessons — The program consists of 12-weekly music lessons, alternating small group lessons and individual lessons each week. Individual lessons reinforce and help personalize what is instructed during group lessons. Lessons are tailored to help older adults with memory challenges learn various instruments, engage in group playing during group lessons, and engage in music appreciation activities. Participants are asked to practice at home in between lessons for 10 minutes per day, 5 times per week, with instruments provided.
  Arms: Music lessons

SUMMARY:
The goal of this pilot clinical trial is to learn if older adults with mild cognitive impairment (MCI) find two music programs equally acceptable. This pilot study will help researchers prepare for a future, large-scale clinical trial to learn if music training can slow cognitive decline and promote emotional well-being in those at risk for Alzheimer's disease and related dementias. The main questions this pilot study aims to answer are:

* Do participants like the music programs?
* Do participants stay enrolled in the study?
* Do participants report perceived benefits of the programs for their emotional well-being or everyday memory?

Participants will:

* Participate in 12-weekly sessions of piano lessons or music lessons, with group and individual lessons alternating each week.
* Have home practice in between lessons, with a keyboard or other instruments provided.
* Keep a diary of their home practice and their mood before and after practice.
* Participate in interviews before and after the 12-week programs.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 60 years
* English-speaking
* Community-dwelling
* Medical diagnosis of MCI by a physician or research diagnostic criteria for MCI, defined by having Montreal Cognitive Assessment (MoCA), with a cutoff of 20- 25 (further adjusted for racial/ethnic differences)
* Capable to consent as identified by the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC)
* No severe psychiatric condition (e.g., bipolar disorder)

Exclusion Criteria:

* Demonstrate musicality knowledge, as assessed by the Musicality Assessment developed by the study team
* Currently participating in a formal music activity (performance, classes, lessons, etc.)
* Major impairment in eyesight or hearing that precludes music reading, hearing, or engagement in the class
* Any difficulty using a keyboard (portable electric piano) due to pain, neuropathy, tremor, or upper finger/hand/limb injury

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent of participants who complete the 12-week program they are randomly assigned to | From enrollment to the end of the program at 12 weeks
  The proportion of participants who complete the program. Feasibility of retention is defined as > 80% of enrolled participants in each group complete at least 10 lesson sessions.

SECONDARY OUTCOMES:
Expectancy of the 12-week program they are randomly assigned to | At enrollment
  This outcome is measured by a 6-item self-reported Credibility/ Expectancy Questionnaire (CEQ) that measure participants' views about the expected efficacy of the 12-week program they are randomly assigned to.
Percent of participants who are approached and consent to the study | At enrollment
  The proportion of participants are approached and consenting to the study. Feasibility of recruitment is defined as > 50% of screened participants consenting to enroll.

OTHER OUTCOMES:
Acceptability of the 12-week program they are randomly assigned to | At enrollment, at the end of the program at 12 weeks
  The acceptability of the program is evaluated through individual interviews conducted before and after the 12-week program. Both interviews are guided by interview guide developed by the research team. The interviews before the program focus on understanding participants' expectations of the program that they are assigned, while the interviews after the program focus on participants' experiences with the program, its design, and areas for improvement.
Satisfaction of the 12-week program they are randomly assigned to | At the end of the program at 12 weeks
  This outcome is measured by a 19-item satisfaction survey developed by the research team. Total scores range from 0 to 80, with higher scores indicating greater satisfaction with the 12-week program to which they are randomly assigned to.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No